CLINICAL TRIAL: NCT03186781
Title: VRC 316: A Phase I Open-Label Clinical Trial To Evaluate Dose, Safety, Tolerability, And Immunogenicity Of An Influenza HA Ferritin Vaccine, Alone Or In Prime-Boost Regimens With An Influenza DNA Vaccine In Healthy Adults
Brief Title: Influenza HA Ferritin Vaccine, Alone or in Prime-Boost Regimens With an Influenza DNA Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 170110; 17-I-0110 (Other: NIH NIAID IRB)
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Influenza
Keywords: Flu Virus; Flu Shot; H2N2; Protein; Immune Response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: HA-F A/Sing (20 mcg), ages 18-47 Yrs (Experimental): HA-F A/Sing injections (20 mcg) administered intramuscularly (IM) by Needle/Syringe (Day 0) in H2-naïve adults (adults with no pre-existing immunity to H2)
  Interventions: Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing)
- Group 2: HA-F A/Sing (60 mcg), ages 18-47 Yrs (Experimental): HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16) in H2-naïve adults (adults with no pre-existing immunity to H2)
  Interventions: Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing)
- Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), ages 18-47 Yrs (Experimental): DNA A/Sing injections (4 mg) administered IM by PharmaJet (Day 0); HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Week 16) in H2-naïve adults (adults with no pre-existing immunity to H2)
  Interventions: Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing); Biological: VRC-FLUDNA082-00-VP (DNA A/Sing)
- Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), ages 52-70 Yrs (Experimental): DNA A/Sing injections (4 mg) administered IM by PharmaJet (Day 0); HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Week 16) in H2-exposed adults (may have some H2 immunity)
  Interventions: Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing); Biological: VRC-FLUDNA082-00-VP (DNA A/Sing)
- Group 4A: HA-F A/Sing (60 mcg), ages 18-47 Yrs (Experimental): HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16) in H2-naïve adults (adults with no pre-existing immunity to H2)
  Interventions: Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing)
- Group 4B: HA-F A/Sing (60 mcg), ages 52-70 Yrs (Experimental): HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16) in H2-exposed adults (may have some H2 immunity)
  Interventions: Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing)

INTERVENTIONS:
Biological: VRC-FLUNPF081-00-VP (HA-F A/Sing) — VRC-FLUNPF081-00-VP (HA-F A/Sing) is an investigational influenza HA ferritin vaccine.
Biological: VRC-FLUDNA082-00-VP (DNA A/Sing) — VRC-FLUDNA082-00-VP (DNA A/Sing) is an investigational influenza plasmid DNA vaccine.
  Arms: Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), ages 18-47 Yrs; Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), ages 52-70 Yrs

SUMMARY:
Background:

Influenza, or "flu", is a very common infectious respiratory disease. Researchers want to develop a vaccine against flu. Vaccines teach the body to fight or prevent an infection. When the body learns to fight an infection, this is called an immune response. In this study, researchers want to test two new vaccines to help the body make an immune response to flu.

Subjects received the vaccine injections in the upper arm muscle. One vaccine, the influenza HA Ferritin vaccine (HA-F A/Sing), was given to all subjects with a needle injection. The other vaccine, influenza DNA vaccine (DNA A/Sing), was given to subjects in Group 3 by a needle-free device that uses high pressure to push the vaccine through the skin and into the muscle.

Objective:

To test the safety and side effects of two new vaccines for prevention of H2 influenza (flu).

Eligibility:

Part I: Healthy adults ages 18-47 born after 1969.

Part II: Healthy adults ages 18-70, but not born in 1966-1969.

Design:

Volunteers were tested for eligibility in a separate screening protocol.

In Part I, all subjects received injections of HA Ferritin vaccine. These subjects were not expected to have H2N2 exposure based on their age and when H2N2 last circulated in the population. Five subjects in Group 1 received one injection of 20 mcg dose vaccine at Day 0 to test if it is safe. Then, five additional subjects in Group 2 received a total of two injections of a 60 mcg dose on Day 0 and 16 weeks later.

In Part II, responses were evaluated from adults born before 1966 who may have prior potential exposure to H2N2 influenza as well as adults similar to those enrolled in Part I who are not expected to have H2N2 exposure. Also, Part II compared responses to 2 different vaccine regimens. Group 3 subjects received a DNA influenza vaccine prime at Day 0 and the HA Ferritin vaccine boost 16 weeks later. Group 4 subjects received the HA Ferritin vaccine 2 times, on Day 0 and 16 weeks later.

DETAILED DESCRIPTION:
Study Design: This is a Phase I open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of VRC-FLUNPF081-00-VP (HA-F A/Sing) vaccine alone or in prime-boost regimens with VRC-FLUDNA082-00-VP (DNA A/Sing) vaccine. The hypotheses are that VRC-FLUNPF081-00-VP and VRC-FLUDNA082-00-VP vaccines are safe, well-tolerated, and induce an immune response to the H2 antigen. The primary objectives are to evaluate the safety and tolerability of two different doses of the HA-F A/Sing vaccine alone and in prime-boost regimens in healthy adults. Secondary objectives are related to the evaluation of the immunogenicity of the HA-F A/Sing and DNA A/Sing vaccines in prime-boost regimens.

Study Products: The investigational HA-F A/Sing vaccine, developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID), is composed of Helicobacter pylori non-haem ferritin with an influenza virus H2 hemagglutinin (HA) insert to form a nanoparticle displaying eight HA trimers from A/Singapore/1/57 (H2N2) influenza.

The investigational DNA A/Sing vaccine, developed by the VRC, NIAID, is composed of a single closed-circular DNA plasmid that encodes the H2 protein of A/Singapore/1/57 influenza.

Subjects: Up to 80 healthy adults ages 18-70 were enrolled; adults born between 1966 and 1969 were excluded from the trial.

Study Plan: Vaccines were administered intramuscularly (IM) in the deltoid muscle. This study has two parts:

Part I evaluated the safety, tolerability, and immunogenicity of 1 or 2 doses of the HA-F A/Sing vaccine in a dose-escalation design. In Group 1, five subjects received a 20 mcg dose of the HA-F A/Sing vaccine via needle and syringe on Day 0. If this dose was assessed as safe and well tolerated, enrollment began for Group 2. In Group 2, five subjects received the higher 60 mcg dose of the HA-F A/Sing vaccine via needle and syringe on Day 0 and Week 16. If this higher dose was assessed as safe, enrollment began for Part II.

Part II evaluated the safety, tolerability, and immunogenicity of HA-F A/Sing vaccine in prime-boost regimens. Subjects were stratified by age and randomized equally into Groups 3 and Group 4. In Group 3, subjects received DNA A/Sing vaccine via a PharmaJet Needle-Free Injector on Day 0 and HA-F A/Sing vaccine via needle and syringe on Week 16. In Group 4, subjects received HA-F A/Sing vaccine via needle and syringe on Day 0 and Week 16.

For Group 1, the protocol required about 8 clinic visits and 1 telephone follow up contact after the injection.

For Group 2, Group 3 and Group 4, the protocol required about 10 clinic visits and 2 telephone follow-up contacts after each injection.

For all Groups, solicited reactogenicity were evaluated using a 7-day diary card. Assessment of vaccine safety included clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

Study Duration: Subjects were evaluated for 40 weeks following the first vaccine administration.

ELIGIBILITY:
INCLUSION CRITERIA:

A subject must meet all of the following criteria:

* Healthy subjects aged 18-70 (excluding subjects born between 1966-1969)
* Based on history and examination, must be in good general health and without history of any of the conditions listed in the exclusion criteria
* Received at least one licensed current seasonal influenza vaccine from 2014 to the present
* Able and willing to complete the informed consent process
* Available for clinic visits for 40 weeks after enrollment
* Willing to have blood samples collected, stored indefinitely, and used for research purposes
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 84 days before enrollment

Laboratory Criteria within 84 days before enrollment:

* White blood cells (WBC) and differential either within institutional normal range or accompanied by the site Principal Investigator (PI) or designee approval
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Platelets = 125,000 - 500,000/mm^3
* Hemoglobin within institutional normal range
* Serum iron either within institutional normal range or accompanied by the site PI or designee approval
* Alanine aminotransferase (ALT) less than or equal to 1.25 times institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) less than or equal to 1.25 times institutional ULN
* Alkaline phosphatase (ALP) less than or equal to 1.1 times institutional ULN
* Total bilirubin within institutional ULN
* Serum creatinine less than or equal to 1.1 times institutional ULN
* Negative for HIV infection by an FDA approved method of detection

Criteria applicable to women of childbearing potential:

* Negative beta-human chorionic gonadotropin (Beta-HCG) pregnancy test (urine or serum) on the day of enrollment
* Agrees to use an effective means of birth control from at least 21 days prior to enrollment through the end of the study

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply:

- Breast-feeding or planning to become pregnant during the study.

Subject has received any of the following substances:

* More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
* Blood products within 16 weeks prior to enrollment
* Live attenuated vaccines within 4 weeks prior to enrollment
* Inactivated vaccines within 2 weeks prior to enrollment.
* Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
* Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Previous H2 influenza investigational vaccine
* Receipt of a licensed influenza vaccine within 6 weeks before trial enrollment

Subject has a history of any of the following clinically significant conditions:

* Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Asthma that is not well controlled
* Diabetes mellitus (type I or II), with the exception of gestational diabetes
* Thyroid disease that is not well controlled
* Idiopathic urticaria within the past year
* Evidence of autoimmune disease or immunodeficiency
* Hypertension that is not well controlled
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* Malignancy that is active or history of malignancy that is likely to recur during the period of the study.
* Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* Guillain-Barre Syndrome
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within 5 years prior to enrollment, a history of suicide plan or attempt
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace L Chen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanekiyo M, Wei CJ, Yassine HM, McTamney PM, Boyington JC, Whittle JR, Rao SS, Kong WP, Wang L, Nabel GJ. Self-assembling influenza nanoparticle vaccines elicit broadly neutralizing H1N1 antibodies. Nature. 2013 Jul 4;499(7456):102-6. doi: 10.1038/nature12202. Epub 2013 May 22. PMID 23698367
- [Background] Yamashita I, Iwahori K, Kumagai S. Ferritin in the field of nanodevices. Biochim Biophys Acta. 2010 Aug;1800(8):846-57. doi: 10.1016/j.bbagen.2010.03.005. Epub 2010 Mar 12. PMID 20227466
- [Background] Nabel GJ, Wei CJ, Ledgerwood JE. Vaccinate for the next H2N2 pandemic now. Nature. 2011 Mar 10;471(7337):157-8. doi: 10.1038/471157a. No abstract available. PMID 21390107
- [Derived] Andrews SF, Raab JE, Gorman J, Gillespie RA, Cheung CSF, Rawi R, Cominsky LY, Boyington JC, Creanga A, Shen CH, Harris DR, Olia AS, Nazzari AF, Zhou T, Houser KV, Chen GL, Mascola JR, Graham BS, Kanekiyo M, Ledgerwood JE, Kwong PD, McDermott AB. A single residue in influenza virus H2 hemagglutinin enhances the breadth of the B cell response elicited by H2 vaccination. Nat Med. 2022 Feb;28(2):373-382. doi: 10.1038/s41591-021-01636-8. Epub 2022 Feb 3. PMID 35115707
- [Derived] Houser KV, Chen GL, Carter C, Crank MC, Nguyen TA, Burgos Florez MC, Berkowitz NM, Mendoza F, Hendel CS, Gordon IJ, Coates EE, Vazquez S, Stein J, Case CL, Lawlor H, Carlton K, Gaudinski MR, Strom L, Hofstetter AR, Liang CJ, Narpala S, Hatcher C, Gillespie RA, Creanga A, Kanekiyo M, Raab JE, Andrews SF, Zhang Y, Yang ES, Wang L, Leung K, Kong WP, Freyn AW, Nachbagauer R, Palese P, Bailer RT, McDermott AB, Koup RA, Gall JG, Arnold F, Mascola JR, Graham BS, Ledgerwood JE; VRC 316 Study Team. Safety and immunogenicity of a ferritin nanoparticle H2 influenza vaccine in healthy adults: a phase 1 trial. Nat Med. 2022 Feb;28(2):383-391. doi: 10.1038/s41591-021-01660-8. Epub 2022 Feb 3. PMID 35115706
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-I-0110.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland.
Period: Overall Study
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs
Started | 5 | 5 | 10 | 10 | 10 | 10
Received First Product Administration | 5 | 5 | 10 | 10 | 10 | 10
Received All Product Administrations | 5 | 5 | 8 (2nd dose not given due to unrelated intercurrent illness (n=1) and lost to follow up (n=1)) | 9 (PI decided not to give 2nd dose to limit variation in environmental exposure to flu between subjects) | 8 (2nd dose not given due to subject decision to withdraw (n=2)) | 9 (PI decided not to give 2nd dose to limit variation in environmental exposure to flu between subjects)
Completed | 5 | 5 | 9 | 10 | 7 | 10
Not Completed | 0 | 0 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Moved from Area | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs | Total
Number analyzed (Participants) | 5 | 5 | 10 | 10 | 10 | 10 | 50
Age, Customized [Count of Participants; unit: Participants]
  18-20 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  21-30 | 2 | 2 | 2 | 0 | 4 | 0 | 10
  31-40 | 3 | 2 | 4 | 0 | 5 | 0 | 14
  41-50 | 0 | 1 | 3 | 0 | 1 | 0 | 5
  51-60 | 0 | 0 | 0 | 6 | 0 | 7 | 13
  61-70 | 0 | 0 | 0 | 4 | 0 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 4 | 6 | 7 | 25
  Male | 4 | 3 | 5 | 6 | 4 | 3 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 1 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1 | 2 | 5 | 9
  White | 4 | 3 | 7 | 7 | 7 | 5 | 33
  More than one race | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Hispanic or Latino | 0 | 1 | 2 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 5 | 4 | 8 | 9 | 10 | 10 | 46
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  18.5-24.9 kg/m^2 | 4 | 3 | 2 | 2 | 6 | 2 | 19
  25.0-29.9 kg/m^2 | 1 | 1 | 8 | 5 | 2 | 5 | 22
  30 kg/m^2 or over | 0 | 1 | 0 | 3 | 2 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Each HA-F A/Sing Product Administration
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after each HA-F A/Sing study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after each HA-F A/Sing product administration, at approximately Week 1 and/or at approximately Week 17
Population: Population included all enrolled subjects who received at least one HA-F A/Sing study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=47). Two subjects in Group 3A and one subject in Group 3B received the prime DNA A/Sing injection but did not receive the boost HA-F A/Sing injection.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence HA-F A/Sing (20 mcg and 60 mcg): HA-F A/Sing dose groups included H2-naïve and H2-exposed adults who received either a single 20 mcg dose of HA-F A/Sing, two doses of 60 mcg HA-F A/Sing 16 weeks apart, or a DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks.
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs | Overall Incidence HA-F A/Sing (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 5 | 8 | 9 | 10 | 10 | 47
Participants
  Pain/Tenderness: None | 4 | 3 | 7 | 9 | 8 | 9 | 40
  Pain/Tenderness: Mild | 1 | 2 | 1 | 0 | 2 | 1 | 7
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 5 | 5 | 8 | 9 | 10 | 10 | 47
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 5 | 5 | 8 | 9 | 10 | 10 | 47
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 4 | 3 | 7 | 9 | 8 | 9 | 40
  Any Local Symptom: Mild | 1 | 2 | 1 | 0 | 2 | 1 | 7
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of DNA A/Sing Product Administration
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after the DNA A/Sing study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after DNA A/Sing product administration, at approximately Week 1
Population: Population included all enrolled subjects who received the DNA A/Sing study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=20).
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence DNA A/Sing (4 mg): DNA A/Sing prime dose groups included H2-naïve and H2-exposed adults who received a DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks.
Arm/Group | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Overall Incidence DNA A/Sing (4 mg)
Number analyzed (Participants) | 10 | 10 | 20
Participants
  Pain/Tenderness: None | 4 | 4 | 8
  Pain/Tenderness: Mild | 6 | 6 | 12
  Pain/Tenderness: Moderate | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0
  Swelling: None | 10 | 10 | 20
  Swelling: Mild | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0
  Redness: None | 10 | 10 | 20
  Redness: Mild | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0
  Any Local Symptom: None | 4 | 4 | 8
  Any Local Symptom: Mild | 6 | 6 | 12
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Each HA-F A/Sing Product Administration
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after each HA-F A/Sing study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after each HA-F A/Sing product administration, at approximately Week 1 and/or at approximately Week 17
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs | Overall Incidence HA-F A/Sing (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 5 | 8 | 9 | 10 | 10 | 47
Participants
  Malaise: None | 4 | 2 | 7 | 7 | 9 | 8 | 37
  Malaise: Mild | 1 | 3 | 1 | 2 | 1 | 2 | 10
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 5 | 3 | 8 | 7 | 7 | 8 | 38
  Myalgia: Mild | 0 | 2 | 0 | 2 | 2 | 2 | 8
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 4 | 1 | 8 | 6 | 8 | 7 | 34
  Headache: Mild | 1 | 4 | 0 | 3 | 2 | 3 | 13
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 5 | 5 | 8 | 9 | 9 | 9 | 45
  Chills: Mild | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 5 | 5 | 8 | 9 | 10 | 9 | 46
  Nausea: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 5 | 5 | 8 | 9 | 9 | 9 | 45
  Joint Pain: Mild | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 5 | 5 | 8 | 9 | 9 | 10 | 46
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Any Systemic Symptom: None | 3 | 1 | 7 | 5 | 7 | 6 | 29
  Any Systemic Symptom: Mild | 2 | 4 | 1 | 4 | 1 | 4 | 16
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 1

4. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of DNA A/Sing Product Administration
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after DNA A/Sing study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after DNA A/Sing product administration, at approximately Week 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Overall Incidence DNA A/Sing (4 mg)
Number analyzed (Participants) | 10 | 10 | 20
Participants
  Malaise: None | 9 | 8 | 17
  Malaise: Mild | 1 | 2 | 3
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Myalgia: None | 9 | 8 | 17
  Myalgia: Mild | 1 | 2 | 3
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Headache: None | 8 | 7 | 15
  Headache: Mild | 2 | 3 | 5
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Chills: None | 10 | 10 | 20
  Chills: Mild | 0 | 0 | 0
  Chills: Moderate | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0
  Nausea: None | 10 | 10 | 20
  Nausea: Mild | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Joint Pain: None | 10 | 10 | 20
  Joint Pain: Mild | 0 | 0 | 0
  Joint Pain: Moderate | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0
  Temperature: None | 10 | 10 | 20
  Temperature: Mild | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0
  Any Systemic Symptom: None | 7 | 6 | 13
  Any Systemic Symptom: Mild | 3 | 4 | 7
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Abnormal Laboratory Measures of Safety
Description: Any abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety laboratory parameters included hematology (hemoglobin, hematocrit, platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil percents/counts) and chemistry (alanine aminotransferase (ALT), alanine aspartate (AST), alkaline phosphate (ALP), creatinine and total bilirubin). Complete blood count (CBC) with differential, total bilirubin, AST, ALT, and ALP results were collected at screening (≤ 84 days before enrollment), Day 0 prior to study product administration (baseline), and at Days 14, 28, 112, 140 and 280. Creatinine results were collected at screening, Day 0 and Day 6. Institutional laboratory normal ranges as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 through Day 280
Population: Population included all enrolled subjects who had laboratory results available at any study visit post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs
Number analyzed (Participants) | 5 | 5 | 10 | 10 | 10 | 10
Participants
  ALP | 0 | 0 | 0 | 0 | 0 | 1
  WBC Count | 1 | 0 | 0 | 1 | 1 | 0
  Hemoglobin | 0 | 2 | 0 | 3 | 4 | 1
  Neutrophil Count | 0 | 0 | 1 | 2 | 1 | 0
  Lymphocyte Count | 0 | 0 | 0 | 2 | 0 | 0
  Eosinophil Count | 0 | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Each HA-F A/Sing Product Administration
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the first study product administration through the visit scheduled for 4 weeks after each study product administration. At other time periods between study product administrations and when greater than 4 weeks after the last study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module), influenza-like illness (ILI) or influenza (reported as a separate outcome) and new chronic medical conditions that required ongoing medical management were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after each HA-F A/Sing product administration, up to Week 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs | Overall Incidence HA-F A/Sing (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 5 | 8 | 9 | 10 | 10 | 47
Participants
  Related to study product | 1 | 0 | 0 | 0 | 1 | 1 | 3
  Unrelated to study product | 3 | 3 | 1 | 3 | 6 | 1 | 17

7. Primary Outcome: Number of Subjects With One or More Unsolicited Non-Serious Adverse Events (AEs) Following DNA A/Sing Product Administration
Description: as for outcome 6
Time Frame: Day 0 through 4 weeks after DNA A/Sing product administration, up to Week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Overall Incidence DNA A/Sing (4 mg)
Number analyzed (Participants) | 10 | 10 | 20
Participants
  Related to study product | 1 | 2 | 3
  Unrelated to study product | 3 | 4 | 7

8. Primary Outcome: Number of Subjects With Influenza or Influenza-like Illness (ILIs) Following HA-F A/Sing Product Administration
Description: Influenza or influenza-like illness (ILI) were recorded in the study database from receipt of the first study product administration through the last study visit.
Time Frame: Day 0 through Day 280
Population: Population included all enrolled subjects who received at least one HA-F A/Sing study injection (N=47). Two subjects in Group 3A and one subject in Group 3B received the prime DNA A/Sing injection but did not receive the boost HA-F A/Sing injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs
Number analyzed (Participants) | 5 | 5 | 8 | 9 | 10 | 10
Participants | 0 | 0 | 1 | 0 | 1 | 0

9. Primary Outcome: Number of Subjects With Influenza or Influenza-like Illness (ILIs) Following DNA A/Sing Product Administration
Description: as for outcome 8
Time Frame: Day 0 through Day 280
Population: Population included all enrolled subjects who received the DNA A/Sing study injection (N=20).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

10. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Following HA-F A/Sing Product Administration
Description: SAEs were recorded from receipt of first study product administration through the last expected study visit at Day 280. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through Day 280
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: HA-F A/Sing (20 mcg), Ages 18-47 Yrs | Group 2: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs | Group 4A: HA-F A/Sing (60 mcg), Ages 18-47 Yrs | Group 4B: HA-F A/Sing (60 mcg), Ages 52-70 Yrs
Number analyzed (Participants) | 5 | 5 | 8 | 9 | 10 | 10
Participants
  Related to study product | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to study product | 0 | 0 | 0 | 1 | 0 | 0

11. Secondary Outcome: Hemagglutination Inhibition Assay (HAI) Geometric Mean Titer (GMT) Against A/Singapore/1/1957 (H2N2) Following the Completion of Each Vaccine Regimen
Description: Hemagglutination inhibition assays (HAI) titers were determined against the homologous H2N2 A/Singapore/1/57 virus, and were summarized using geometric mean titers (GMTs). Negative samples were reported and GMTs were calculated using half the limit of detection. H2-naïve (ages 18-47 years) and H2-exposed (ages 52-70 years) subjects received either a single dose of 20 mcg HA-F A/Sing (H2-naïve), two doses of 60 mcg HA-F A/Sing 16 weeks apart (H2-naïve and H2-exposed), or a 4 mg DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks (H2-naïve and H2-exposed).
Time Frame: Four weeks after the first dose for groups that received a single vaccination, at Week 4 or two weeks after the second dose for groups that received two vaccinations, at Week 18
Population: Overall number analyzed includes the H2-naïve adults (adults with no pre-existing immunity to H2) and H2-exposed adults (may have some H2 immunity). The H2-naïve and H2-exposed number analyzed rows reflect the number of subjects analyzed in each group.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- HA-F A/Sing (20 mcg), Ages 18-47 Yrs: HA-F A/Sing injections (20 mcg) administered intramuscularly (IM) by Needle/Syringe (Day 0) in H2-naïve adults (adults with no pre-existing immunity to H2)
  VRC-FLUNPF081-00-VP (HA-F A/Sing): VRC-FLUNPF081-00-VP (HA-F A/Sing) is an investigational influenza HA ferritin vaccine.
- HA-F A/Sing (60 mcg), Ages 18-47 and 52-70 Yrs: HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16) in H2-naïve adults (adults with no pre-existing immunity to H2) and H2-exposed adults (may have some H2 immunity)
  VRC-FLUNPF081-00-VP (HA-F A/Sing): VRC-FLUNPF081-00-VP (HA-F A/Sing) is an investigational influenza HA ferritin vaccine.
- DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 and 52-70 Yrs: DNA A/Sing injections (4 mg) administered IM by PharmaJet (Day 0); HA-F A/Sing injections (60 mcg) administered IM by Needle/Syringe (Week 16) in H2-naïve adults (adults with no pre-existing immunity to H2) and H2-exposed adults (may have some H2 immunity)
Arm/Group | HA-F A/Sing (20 mcg), Ages 18-47 Yrs | HA-F A/Sing (60 mcg), Ages 18-47 and 52-70 Yrs | DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 and 52-70 Yrs
Number analyzed (Participants) | 5 | 22 | 18
titer
  H2-naïve: number analyzed (Participants) | 5 | 13 | 9
  H2-naïve | NA [NA to NA] — Values are below lower limit of quantitation for the assay (GMT was less than 10) | 24 [14 to 40] | 89 [28 to 282]
  H2-exposed: number analyzed (Participants) | 0 | 9 | 9
  H2-exposed |  | 64 [22 to 189] | 113 [71 to 179]

12. Secondary Outcome: Pseudoviral Neutralization Assay Geometric Mean Titer (GMT) Against A/Singapore/1/1957 (H2N2) Following the Completion of Each Vaccine Regimen
Description: Pseudoviral neutralization antibody titers were determined against the homologous H2N2 A/Singapore/1/57 virus, and were summarized using geometric mean 50% inhibitory concentration (IC50). Negative samples were reported and IC50 titers were calculated using half the limit of detection. H2-naïve (ages 18-47 years) and H2-exposed (ages 52-70 years) subjects received either a single dose of 20 mcg HA-F A/Sing (H2-naïve), two doses of 60 mcg HA-F A/Sing 16 weeks apart (H2-naïve and H2-exposed), or a 4 mg DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks (H2-naïve and H2-exposed).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | HA-F A/Sing (20 mcg), Ages 18-47 Yrs | HA-F A/Sing (60 mcg), Ages 18-47 and 52-70 Yrs | DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 and 52-70 Yrs
Number analyzed (Participants) | 5 | 22 | 18
titer
  H2-naïve: number analyzed (Participants) | 5 | 13 | 9
  H2-naïve | 127 [65 to 251] | 844 [382 to 1868] | 2723 [551 to 13466]
  H2-exposed: number analyzed (Participants) | 0 | 9 | 9
  H2-exposed |  | 1279 [351 to 4665] | 2718 [1041 to 7099]

13. Secondary Outcome: Seroconversion Rate Following the Completion of Each Vaccine Regimen
Description: Seroconversion rate: the proportion of subjects achieving seroconversion in hemagglutination inhibition assay (HAI) antibody titer. Seroconversion rates for HAI were summarized as the proportion of individuals in each group experiencing a positive response, defined per the FDA criteria of positivity as either a baseline titer of less than 1:10 and a post vaccination titer of 1:40 or more or a baseline titer of 1:10 or more and a minimum four-fold rise after vaccination. H2-naïve (ages 18-47 years) and H2-exposed (ages 52-70 years) subjects received either a single dose of 20 mcg HA-F A/Sing (H2-naïve), two doses of 60 mcg HA-F A/Sing 16 weeks apart (H2-naïve and H2-exposed), or a 4 mg DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks (H2-naïve and H2-exposed).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HA-F A/Sing (20 mcg), Ages 18-47 Yrs | HA-F A/Sing (60 mcg), Ages 18-47 and 52-70 Yrs | DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 and 52-70 Yrs
Number analyzed (Participants) | 5 | 22 | 18
percentage of participants
  H2-naïve: number analyzed (Participants) | 5 | 13 | 9
  H2-naïve | 0 [0 to 52] | 31 [9.1 to 61] | 78 [40 to 97]
  H2-exposed: number analyzed (Participants) | 0 | 9 | 9
  H2-exposed |  | 56 [21 to 86] | 89 [52 to 100]

14. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Following DNA A/Sing Product Administration
Description: as for outcome 10
Time Frame: Day 0 through Day 280
Population: Population included all enrolled subjects who received the DNA A/Sing study injection (N=20).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3A: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 18-47 Yrs | Group 3B: DNA A/Sing(4 mg)-HA-F A/Sing(60 mcg), Ages 52-70 Yrs
Number analyzed (Participants) | 10 | 10
Participants
  Related to study product | 0 | 0
  Unrelated to study product | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study injection. Unsolicited AEs were recorded from receipt of the first study injection through the visit scheduled 4 weeks after each study injection. At other time periods between injections and when greater than 4 weeks after the last injection, only serious AEs, influenza or influenza-like illness (ILI) and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: The overall Arms/Groups summarize AEs collected after each product administration separately and grouped by the study product and dose, including the groups in which 2 different products were administered. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of subjects reporting the event. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Groups:
- Overall Incidence HA-F A/Sing (20 mcg): HA-F A/Sing (20 mcg) dose group included H2-naïve (ages 18-47 years) adults who received a single 20 mcg dose of HA-F A/Sing.
  Population included all enrolled subjects who received a HA-F A/Sing (20 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=5).
  VRC-FLUNPF081-00-VP (HA-F A/Sing): VRC-FLUNPF081-00-VP (HA-F A/Sing) is an investigational influenza HA ferritin vaccine.
- Overall Incidence HA-F A/Sing (60 mcg): HA-F A/Sing (60 mcg) dose groups included H2-naïve (ages 18-47 years) and H2-exposed (ages 52-70 years) adults who received either two doses of 60 mcg HA-F A/Sing 16 weeks apart, or a DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks.
  Population included all enrolled subjects who received at least one HA-F A/Sing (60 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=42). Two subjects in Group 3A and one subject in Group 3B received the prime DNA A/Sing injection but did not receive the boost HA-F A/Sing injection.
  VRC-FLUNPF081-00-VP (HA-F A/Sing): VRC-FLUNPF081-00-VP (HA-F A/Sing) is an investigational influenza HA ferritin vaccine.
  VRC-FLUDNA082-00-VP (DNA A/Sing): VRC-FLUDNA082-00-VP (DNA A/Sing) is an investigational influenza plasmid DNA vaccine.
- Overall Incidence DNA A/Sing (4 mg): DNA A/Sing prime dose groups included H2-naïve (ages 18-47 years) and H2-exposed (ages 52-70 years) adults who received a DNA A/Sing prime followed by a single 60 mcg HA-F A/Sing boost at 16 weeks.
  Population included all enrolled subjects who received the DNA A/Sing study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=20).
  VRC-FLUDNA082-00-VP (DNA A/Sing): VRC-FLUDNA082-00-VP (DNA A/Sing) is an investigational influenza plasmid DNA vaccine.
Arm/Group | Overall Incidence HA-F A/Sing (20 mcg) | Overall Incidence HA-F A/Sing (60 mcg) | Overall Incidence DNA A/Sing (4 mg)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/42 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/42 | 0/20
Other Adverse Events (participants affected / at risk) | 4/5 | 21/42 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Incidence HA-F A/Sing (20 mcg) (N=5) | Overall Incidence HA-F A/Sing (60 mcg) (N=42) | Overall Incidence DNA A/Sing (4 mg) (N=20)
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Incidence HA-F A/Sing (20 mcg) (N=5) | Overall Incidence HA-F A/Sing (60 mcg) (N=42) | Overall Incidence DNA A/Sing (4 mg) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 8 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 4
Hypertension (Vascular disorders) | 0 | 0 | 1
Administration site pain (General disorders) | 1 | 6 | 12
Malaise (General disorders) | 1 | 9 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 9 | 3
Headache (Nervous system disorders) | 1 | 12 | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03186781/Prot_SAP_ICF_000.pdf